CLINICAL TRIAL: NCT05966766
Title: Estimating the Effective Dose of Music Duration for Anxiety Reduction Prior to Cesarean Delivery
Brief Title: Dosing Music for Anxiety Reduction in Parturients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00003958
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Results first posted 2025-05-30 (Actual); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mozart (Active Comparator): Subjects in this arm will listen to music from a list of pre-selected pieces by Mozart that have been previously shown to have beneficial effects on anxiety.
  Interventions: Other: Mozart selections
- Patient preference (Active Comparator): Subjects in this arm will listen to music from a list of pre-selected pieces of their own choosing.
  Interventions: Other: Patient-preferred music selections

INTERVENTIONS:
Other: Mozart selections — Music will be played from a speaker connected to a media-playing device for participants to listen to for set durations of time. Music will be selections by Mozart of previously studied and shown to reduce anxiety.
  Arms: Mozart
Other: Patient-preferred music selections — Music will be played from a speaker connected to a media-playing device for participants to listen to for set durations of time. Music will be selections of patient choice.
  Arms: Patient preference

SUMMARY:
This is a clinical study that aims to determine the effective dose of music listening duration that is required to reduce anxiety in patients awaiting scheduled cesarean section. It will also compare types of music to accomplish this goal, both of which have been shown effective in prior studies. Methods will involve enrolling and playing music for patients awaiting scheduled C-section, and scoring their anxiety with pre- and post-music questionnaires. Music duration for each subject will be predetermined, and analysis of response will be performed to determine the effective dose 95%, or dose at which 95% of subjects should have a positive response.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Planning on scheduled cesarean section or non-emergent unscheduled cesarean section
* Able to provide informed consent
* American Society of Anaesthesiologists (ASA) physical status score of II-III

Exclusion Criteria:

* Patient refusal
* Impaired hearing
* Patient is taking at least one anxiolytic medication daily at baseline
* No anxiety (a score of 0, on a scale of 0-10, of pre-music exposure anxiety) after consent is given
* ASA IV or higher

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-12-07 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dan Drzymalski, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mozart | Patient Preference
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of individuals grouped by intervention received.
Groups:
- Mozart: Subjects in this arm listened to music from a list of pre-selected pieces by Mozart that have been previously shown to have beneficial effects on anxiety.
- Patient Preference: Subjects in this arm listened to music from a list of pre-selected pieces of their own choosing.
- Total: Total of all reporting groups
Arm/Group | Mozart | Patient Preference | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.7 (5.4) | 33.5 (4.9) | 33.0 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 16 | 16 | 32
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 5 | 13
  White | 10 | 12 | 22
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Gestational age [Mean (Standard Deviation); unit: Weeks] | 38.6 (0.8) | 38.6 (0.9) | 38.6 (0.9)
Gravidity [Mean (Standard Deviation); unit: Pregnancies] | 2.4 (1) | 3.6 (1.3) | 3 (2.2)
Parity [Mean (Standard Deviation); unit: Births] | 1.1 (0.8) | 1.3 (1.4) | 1.2 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Anxiety Score
Description: Verbally rated anxiety on numeric rating scale (NRS) of 0-10, before and after intervention. A rating of 0 meant the patient had no anxiety, while a rating of 10 meant the patient had the worst anxiety possible. Must have been at least a 1-point decrease between pre- and post-intervention scores to be considered a positive response, larger decrease meant a better outcome.
Time Frame: 4-8 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mozart | Patient Preference
Number analyzed (Participants) | 20 | 20
score on a scale
  Before | 5.9 (2.6) | 6.1 (2.3)
  After | 3.6 (2.3) | 3.1 (2.4)

2. Secondary Outcome: STAI
Description: 6-question abbreviated state-trait anxiety inventory (STAI) questions asked and scored on a 6-24 point scale (higher is more anxiety) for before and after intervention. Decrease in score after intervention was considered a positive response, with larger decreases indicating better responses.
Time Frame: 4-8 minutes
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mozart | Patient Preference
Number analyzed (Participants) | 20 | 20
score on a scale
  Before | 12.7 (4.3) | 14.4 (4.1)
  After | 10.3 (3.2) | 10.8 (3.2)

ADVERSE EVENTS:
Time Frame: 1 day
Arm/Group | Mozart | Patient Preference
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

LIMITATIONS AND CAVEATS:
Minimum required number of participants recruited was achieved. Larger sample sizes may have yielded results of stronger statistical significance.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-31): https://cdn.clinicaltrials.gov/large-docs/66/NCT05966766/Prot_SAP_000.pdf